CLINICAL TRIAL: NCT06880120
Title: Improvement of Diagnostic Accuracy of Seismocardiography and Gyrocardiography for Non-Invasive Coronary Artery Disease Diagnosis: A Comparison With Coronary Artery Calcium Computed Tomography, Coronary Computed Tomography Angiography, and Invasive Coronary Angiography
Brief Title: Diagnostic Accuracy Of Seismocardiography for Coronary Artery Disease
Acronym: HF-CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Force Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UZ-1-16-02-388-19
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease (CAD) (E.G., Angina, Myocardial Infarction, and Atherosclerotic Heart Disease (ASHD))
Keywords: coronary artery disease; Seismocardiography; CardioClin
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Infarction | interventions — Diagnostic Techniques and Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of the CardioClin SCG/GCG Device for Coronary Artery Disease Diagnosis (Experimental): Participants in this arm will undergo seismocardiography (SCG) and gyrocardiography (GCG) testing using the CardioClin device, a non-invasive diagnostic tool designed to assess coronary artery disease (CAD). The device uses high-precision accelerometers and gyroscopic sensors to measure the mechanical vibrations of the heart.
  All participants are already scheduled for standard diagnostic procedures such as coronary artery calcium computed tomography (CAC-CT), coronary computed tomography angiography (CCTA), or invasive coronary angiography (ICA). SCG/GCG testing will be performed before these standard procedures, with measurements taken in both supine and sitting positions.
  The goal is to compare the diagnostic accuracy of CardioClin SCG/GCG recordings against traditional imaging methods to assess its potential as a non-invasive alternative for CAD detection.
  Interventions: Device: Seismocardiography (SCG) and Gyrocardiography (GCG) Diagnostic Testing

INTERVENTIONS:
Device: Seismocardiography (SCG) and Gyrocardiography (GCG) Diagnostic Testing — This intervention involves the use of Seismocardiography (SCG) and Gyrocardiography (GCG) Diagnostic Testing, a non-invasive technique that records mechanical vibrations of the chest caused by heart activity using high-precision accelerometers and gyroscopes. Unlike traditional imaging techniques such as coronary artery calcium computed tomography (CAC-CT), coronary computed tomography angiography (CCTA), and invasive coronary angiography (ICA), this method does not require radiation exposure (unlike CAC-CT and CCTA), is completely non-invasive and does not require contrast agents (unlike ICA), and provides real-time cardiac mechanical activity measurements rather than anatomical imaging.

SUMMARY:
This study aims to evaluate a new, non-invasive method for detecting coronary artery disease (CAD) using seismocardiography (SCG) and gyrocardiography (GCG). These techniques measure small vibrations on the chest caused by the heartbeat using highly sensitive sensors. The goal is to determine whether this method, using the CardioClin device, can accurately detect CAD compared to standard tests like coronary calcium scans (CAC-CT), CT angiography (CCTA), and invasive coronary angiography (ICA).

Patients who are already scheduled for one of these standard tests will also undergo SCG/GCG testing. The study will compare results to see if the new method provides a reliable, cost-effective, and radiation-free alternative for diagnosing CAD.

This research could help improve early detection of heart disease without the need for invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Suspected CAD, based on clinical evaluation.
* Able to provide informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Presence of implanted cardiac devices (e.g., pacemakers, implantable cardioverter defibrillators) that may interfere with SCG/GCG signal acquisition.
* Severe arrhythmias that may affect signal interpretation.
* Inability to maintain required testing positions (supine and sitting).
* Medical conditions preventing informed consent (e.g., severe cognitive impairment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1534 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-11-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of SCG/GCG for Coronary Artery Disease (CAD) Detection | Baseline (Day 1, before standard diagnostic procedures).
  The ability of Seismocardiography (SCG) and Gyrocardiography (GCG) testing to accurately detect coronary artery disease (CAD) compared to standard diagnostic methods (CAC-CT, CCTA, ICA).

CONTACTS AND LOCATIONS:
Locations (1):
- Republic Specialized Scientific-Practical Medical Center of Cardiology (RSPCMCC), Tashkent, Uzbekistan